CLINICAL TRIAL: NCT03982433
Title: Internet-based Video-conferencing to Address Alcohol Use and Pain Among Heavy Drinkers in HIV-care
Brief Title: Internet-based Videoconferencing to Address Alcohol Use and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4546; UH2AA026192 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-06-11 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain; Alcohol Use, Unspecified
Keywords: HIV
MeSH Terms: conditions — Chronic Pain; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants all undergo assessment and intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): participants all receive the intervention
  Interventions: Behavioral: Motivation and Cognitive Behavioral Management for Alcohol and Pain

INTERVENTIONS:
Behavioral: Motivation and Cognitive Behavioral Management for Alcohol and Pain — Behavioral intervention that includes motivational, cognitive, and behavioral intervention strategies to reduce heavy drinking and chronic pain interference

SUMMARY:
This research seeks to develop a novel, integrated behavioral approach to reduce heavy drinking and chronic pain among patients in HIV-care delivered via internet-based videoconferencing. This first open trial pilot study seeks to recruit patients in the clinic through posted flyers, cards and physician referral.

DETAILED DESCRIPTION:
This study seeks to develop an integrated, behavioral video telehealth approach to address pain and heavy alcohol use among patients living with HIV and determine its feasibility and acceptability. Through an open pilot trial, this phase of this project will deliver an integrated alcohol-pain behavioral intervention to people living with HIV/AIDS (PLWHA) through videoconferencing. Intervention evaluation outcomes for this initial phase will include reduction of standard number of drinks per week, reduction in heavy drinking days, reduction of chronic pain severity and interference, ratings of patient satisfaction with treatment, and rate of treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* engaged in HIV care, heavy drinking by more than 7/14 drinks per week (women/men) or by single episode of 4/5 (women/men), chronic (at least 3 months duration) moderate or greater (4 or more on the severity scale of the Brief Pain Inventory (BPI) non-cancer related pain.

Exclusion Criteria:

* psychoactive medication for pain or alcohol use for few than 2 months
* history of bipolar disorder, schizophrenia, other psychotic disorder
* current suicidal intent
* prior history of alcohol withdrawal related seizures or delirium tremens
* current behavioral treatment for pain or alcohol use
* any scheduled surgery within next 6 months or acute life-threatening illness that requires treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor P Palfai, PhD, Principal Investigator — Boston University
Locations (1):
- General Clinical Research Unit, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palfai TP, Kratzer MPL, Taylor JL, Otis JD, Winter MR. Addressing Pain and Heavy Drinking among Patients in HIV-Care: A Pilot Study of an Integrated Telehealth Intervention. AIDS Behav. 2025 Jun;29(6):1930-1943. doi: 10.1007/s10461-025-04660-8. Epub 2025 Feb 25. PMID 39998790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from medical clinic and ongoing cohort
Groups:
- Intervention: 8 participants assigned to receive the intervention
  Motivation and Cognitive Behavioral Management for Alcohol and Pain: Behavioral intervention that includes motivational, cognitive, and behavioral intervention strategies to reduce heavy drinking and chronic pain interference
Period: Overall Study
Arm/Group | Intervention
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Brief Pain Inventory (BPI) [Median (Standard Deviation); unit: units on a scale] — BPI consists of 11-point scale items that reflect pain severity and pain interference
  Average pain severity in the past 7-days is measures with a single 11-point scale where "0" is best and "10" is worst.
  Pain interference is measured as the mean of 7-items, each also rated on a 11-point scale where "0" is best and "10 is worst"
  Scales range from 0 - 10
  units on a scale
    pain severity | 5.5 (1.52)
    pain interference | 4.5 (2.24)
Heavy Drinking Episodes [Median (Standard Deviation); unit: episodes] — Calendar-based measure of the number of heavy drinking episodes in the past 30 days.
  episodes | 5.5 (5.62)
Drinks/week from Timeline FollowBack [Median (Standard Deviation); unit: drinks/week] — Calendar-based measure of the number of drinks per week over the prior month. The average drinks per week is computed by (Total drinks/4.28)
  drinks/week | 36.50 (18.43)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Pain Severity
Description: BPI consists of 11-point scale items that reflect pain severity and pain interference Average pain severity in the past 7-days is measures with a single 11-point scale where "0" is best and "10" is worst.
  Pain interference is measures as the mean of 7-items, each also rated on a 11-point scale where "0" is best and "10 is worst" Scales range from 0 - 10
Time Frame: past 7 days
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Intervention: 8 participants all receive the intervention
  Motivation and Cognitive Behavioral Management for Alcohol and Pain: Behavioral intervention that includes motivational, cognitive, and behavioral intervention strategies to reduce heavy drinking and chronic pain interference
Arm/Group | Intervention
Number analyzed (Participants) | 7
units on a scale | 5.0 (2.58)

2. Primary Outcome: Brief Pain Inventory Pain Interference
Description: BPI consists of 11-point scale items that reflect pain severity and pain interference
  Pain interference is measured as the mean of 7-items, each rated on a 11-point scale where "0" is best and "10 is worst" Scales range from 0 - 10
Time Frame: past 7 days
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
units on a scale | 2.43 (2.68)

3. Primary Outcome: Alcohol Time Line Follow Back...Heavy Drinking Episodes
Description: number of heavy drinking episodes in the past 30 days
Time Frame: past 30 days
Measure: Median (Standard Deviation); unit: number of episodes
Arm/Group | Intervention
Number analyzed (Participants) | 7
number of episodes | 2.0 (4.34)

4. Primary Outcome: Alcohol Time Line Follow Back...Average Drinks Per Week
Description: average number of drinks per week in the past 30 days (total number of drinks 30 days/4.28)
Time Frame: past 30 days
Measure: Median (Standard Deviation); unit: drinks/week
Arm/Group | Intervention
Number analyzed (Participants) | 7
drinks/week | 13 (21.57)

5. Primary Outcome: Client Satisfaction Questionnaire-8 [Modified]
Description: Evaluative ratings of the intervention received. Eight Likert-scale items regarding different components of treatment satisfaction are rated from 1-4. Some items are reversed scored and then they are summed so that higher scores reflect higher satisfaction with treatment.
  The possible range of scores is 8-32.
Time Frame: past 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
units on a scale | 29.29 (2.29)

6. Primary Outcome: Perceptions of Treatment Questionnaire
Description: Participants were asked about their experiences with different facets of the intervention using items that were scored from 0 - 8 with higher scores reflecting greater satisfaction with the treatment components.
Time Frame: past 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
units on a scale | 7.04 (1.15)

7. Secondary Outcome: Goal Systems Assessment Battery-Pain
Description: Ratings self-regulatory capacities related to pain. Participants rate their perceived self-regulatory skills related to pain management using 5-point Likert scale items. There are 4 subscales for each of the dimensions of self-regulation assessed; planning, monitoring, self-efficacy, and value about the behavior change goal. A mean scale score is taken for each subscale. The range for each subscale is 0-4. Higher scores reflect better outcomes.
Time Frame: past 30 days
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
score on a scale
  Pain-Value | 3.25 (0.70)
  Pain-Self-efficacy | 3.0 (0.84)
  Pain-Monitoring | 3.0 (0.92)
  Pain-Planning | 2.75 (0.89)

8. Secondary Outcome: Goal Systems Assessment Battery-Alcohol
Description: Ratings self-regulatory capacities related to moderating alcohol use. Participants rate their perceived self-regulatory skills related to pain management using 5-point Likert scale items. There are 4 subscales for each of the dimensions of self-regulation assessed; planning, monitoring, self-efficacy, and value about the behavior change goal. A mean scale score is taken for each subscale. The range for each subscale is 0-4. Higher scores reflect better outcomes.
Time Frame: past 30 days
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
units on a scale
  Alcohol-Value | 3.0 (0.87)
  Alcohol-Self-efficacy | 3.0 (0.71)
  Alcohol-Monitoring | 2.75 (0.82)
  Alcohol-Planning | 2.75 (0.89)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: no difference
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT03982433/Prot_SAP_000.pdf